CLINICAL TRIAL: NCT07029113
Title: Effects of Task-Oriented Training and Mulligan Mobilization on Hand Function, Pain and Quality of Life in Patients With Rheumatoid Arthritis: A Randomized Controlled Study
Brief Title: Effects of Task-Oriented Training and Mulligan Mobilization on Hand Function, Pain and Quality of Life in Patients With Rheumatoid Arthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kirsehir Ahi Evran Universitesi (Other)
Responsible Party: Principal Investigator, Mehmet CANLI, Lecturer, Kirsehir Ahi Evran Universitesi
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 43834581758"
Record Dates: First submitted 2025-06-08; First posted 2025-06-19 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-06

CONDITIONS: Rheumatic Arthritis
Keywords: Rheumatic arthritis; Treatment; Mobilization
MeSH Terms: conditions — Rheumatic Fever

STUDY DESIGN:
Intervention Model Description: Randomized controlled trials
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Conventional Group (Experimental): Conventional Group, the patients performed passive range of motion (PROM) exercises, mobilization of MCP, PIP and distal interphalangeal (DIP) joints and isometric exercises. While PROM and isometric exercises were applied in 30 repetitions, joint mobilizations were performed by the therapist with moderate severity in the form of anteroposterior and mediolateral gliding.
  Interventions: Other: Conventional treatment
- Mulligan Mobilization Group (Experimental): In the Mulligan mobilisation group, the therapist will apply a dorsal shift from the distal radius to the carpal bones and the patient will simultaneously extend the wrist. It is essential that the movement is painless; if any pain occurs during mobilisation, the direction or technique will be re-evaluated. This application will be performed in 8-10 repetitions and the frequency of the session will be planned according to the patient's symptoms.
  Interventions: Other: Mulligan mobilization; Other: Conventional treatment
- Task-Oriented Training Group (Experimental): In addition to MCP, PIP, DIP joint mobilisation and isometric exercises, the task-oriented training group will perform 30 repetitions of face washing, using a fork, drinking water with a glass, sitting and wearing a t-shirt exercises.
  Interventions: Other: Task-oriented trainig; Other: Conventional treatment

INTERVENTIONS:
Other: Task-oriented trainig — In addition to MCP, PIP, DIP joint mobilisation and isometric exercises, the task-oriented training group will perform 30 repetitions of face washing, using a fork, drinking water with a glass, sitting and wearing a t-shirt exercises.
  Arms: Task-Oriented Training Group
Other: Mulligan mobilization — In patients included in the Mulligan mobilisation group, the therapist will apply a dorsal shift from the distal radius to the carpal bones and the patient simultaneously extends the wrist. It is essential that the movement is painless; if any pain occurs during mobilisation, the direction or technique is re-evaluated. This application is performed in 8-10 repetitions and the frequency of the session is planned according to the patient's symptoms.
  Arms: Mulligan Mobilization Group
Other: Conventional treatment — Passive range of motion exercises, metacarpopalangeal, proximal interphalangeal and distal interphalangeal joint mobilisation and isometric exercises will be applied. Isometric exercises will be performed as 30 repetitions, while joint mobilisations will be performed by the therapist as moderate anteroposterior and mediolateral shifts.

SUMMARY:
Rheumatoid arthritis (RA) is a chronic and progressive inflammatory disease that frequently affects the hand joints. Over time, this disease leads to joint deformities, pain, decreased muscle strength and severe impairment in hand function. Functions such as independence in activities of daily living, hand skills and grip strength may be significantly limited in individuals with RA. Although hand rehabilitation is an important component of RA management, there is still a need for research on effective intervention strategies.

DETAILED DESCRIPTION:
Rheumatoid arthritis (RA) is a chronic and progressive inflammatory disease that frequently affects the hand joints. Over time, this disease leads to joint deformities, pain, decreased muscle strength and severe impairment in hand function. Functions such as independence in activities of daily living, hand skills and grip strength may be significantly limited in individuals with RA. Although hand rehabilitation is an important component of RA management, there is still a need for research on effective intervention strategies.

Conventional exercises are basic applications to maintain range of motion, muscle strength and endurance. However, these approaches may have limited effects on improving hand function. In recent years, methods such as task-oriented training and Mulligan mobilisation have gained attention for their potential to improve neuromotor control, hand dexterity and pain. Task-oriented training promotes motor learning through functional tasks, while Mulligan mobilisation aims to increase mobility through pain-free passive-joint mobilisation techniques. The effects of these two methods, separately or in combination, on hand function, pain level and quality of life in individuals with RA have not been adequately investigated.

The aim of this study was to investigate the effects of task-focused training and Mulligan mobilisation on hand function, grip strength, dexterity, pain, activities of daily living and quality of life in individuals with RA.

ELIGIBILITY:
Inclusion Criteria:

* Followed for at least one year for the diagnosis of Rheumatoid Arthritis, aged between 30 and 65,
* Have the cognitive capacity to understand and follow the instructions given,
* Has not undergone upper extremity surgery for orthopaedic, neurological or other reasons
* Participants with functional capacity class I-II

Exclusion Criteria:

* Severe pain as assessed by Visual Analogue Scale (VAS) (VAS >7),
* Declaring the intention to withdraw from the study without giving any reason,
* Having a major psychiatric disorder such as schizophrenia or major depression,
* Having cardiovascular diseases such as coronary artery disease, history of myocardial infarction, angina, stroke, uncontrolled hypertension, chronic obstructive pulmonary disease (COPD)

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2025-07-01 (Actual); Primary Completion 2025-11-08 (Actual); Study Completion 2025-11-08 (Actual)

PRIMARY OUTCOMES:
Evaluation of Hand Grip Strength | 5 week
  Hand grip strength of the participants was measured with a hand dynamometer (Takei Scientific Instruments Co., Ltd., Japan). During the test application, the standard positioning rules determined by the American Association of Hand Therapists will be followed. Accordingly, the participant will be ensured to be in an upright sitting position and the consistency of the measurements will be maintained by not allowing the arms to be supported.

SECONDARY OUTCOMES:
Evaluation of Hand Functions | 5 week
  Nine-Hole Peg Test and Duruöz Hand Index will be used for the evaluation of hand functions. The Nine-Hole Peg Test is a practical and rapidly applicable manual skill measurement method with scientifically proven validity and reliability. The Duruöz Hand Index was first developed in 1996 to assess hand function in patients with Rheumatoid Arthritis. Since then, it has been shown to be valid and reliable in a wide range of upper extremity conditions. It consists of 18 questions.
Evaluation of Pain Severity | 5 week
  The pain intensity of the participants will be evaluated with the McGill-Melzack Pain Questionnaire.
Assessment of Quality of Life | 5 week
  The Rheumatoid Arthritis Quality of Life Questionnaire will be used to assess patient-specific symptoms and the impact of the disease on life. The Rheumatoid Arthritis Quality of Life Scale is a unique 30-item quality of life assessment tool for RA patients developed in parallel studies in the UK and the Netherlands.
Disease Activity | 5 week
  The Disease Activity Score-28 (DAS-28) is a widely used measure in clinical settings to assess disease activity in individuals with RA. The score is derived from the number of swollen and tender joints in the patient's 28 joints, the acute-phase reactants (erythrocyte sedimentation rate, ESR, or CRP), and a 0-100 mm visual analog scale (VAS) score that reflects the patient's overall health status. The DAS-28 score categorizes disease activity as low, moderate, or high.

CONTACTS AND LOCATIONS:
Overall Officials: Mehmet CANLI, PhD., Study Director — Kirsehir Ahi Evran Universitesi
Locations (1):
- Kırşehir Ahi Evran University, Kırşehir, Kırşehir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No